CLINICAL TRIAL: NCT02396680
Title: An Observational Follow-On Field Study to Evaluate the Continued Efficacy and Safety of Ragweed-SPIRE Treatment in Ragweed Allergic Subjects Approximately One Year After the Completion of Treatment
Brief Title: Ragweed-SPIRE Follow-On Study
Status: Completed | Type: Observational
Sponsor: Circassia Limited (Industry)
Collaborators: Adiga Life Sciences, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: TR006A
Record Dates: First submitted 2015-03-19; First posted 2015-03-24 (Estimated); Last update posted 2016-03-23 (Estimated); Status verified 2016-03

CONDITIONS: Rhinoconjunctivitis; Ragweed Allergy
Keywords: Ragweed Allergy; Rhinoconjunctivitis; Immunotherapy; Ragweed-SPIRE

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- TR006 Subjects: Subjects that have previously been randomised into study TR006

SUMMARY:
The purpose of this study is to determine the efficacy of Ragweed-SPIRE 12 months after the initial dose.

ELIGIBILITY:
Inclusion Criteria:

° Previously randomised into and completed at least 6 of 8 treatment visits in Study TR006

Exclusion Criteria:

* Subject or Investigator have been informed of treatment received in Study TR006
* Subjects with significant allergy to animal dander
* Any allergen immunotherapy since completing Study TR006 or use of prohibited therapies
* History of recurrent acute sinusitis or chronic sinusitis
* Received treatment with an investigational drug within 4 weeks of Screening
* Unable to understand study requirements or unable to communicate clearly with Investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who completed at least 6 of 8 treatment visits in Study TR006
Sampling Method: Non-Probability Sample
Enrollment: 249 (Actual)
Dates: Start 2015-04; Primary Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Total Rhinoconjunctivitis Symptom Score | Approximately 12 months after first dose in TR006

SECONDARY OUTCOMES:
Rescue Medication Score | Approximately 12 months after first dose in TR006
Patient Global Assessment | Approximately 12 months after first dose in TR006
Skin Prick Test | Approximately 12 months after first dose in TR006
Immunoglobulin E Test | Approximately 12 months after first dose in TR006

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - Kanata Allergy Services, Kanata, Ontario
  - Inflamax Research, Mississauga, Ontario
  - Windsor Allergy Asthma Associates, Windsor, Ontario